CLINICAL TRIAL: NCT01839409
Title: Biological Rhythms and Vestibular System
Acronym: REHAB_Rn'V
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-A001359-32; N° 11P03919 / N°11P03921 (Other Grant/Funding Number: CRBN)
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Unspecified Disorder of Vestibular Function, Bilateral
Keywords: Circadian Rhythm; Exercise; Reflex, Vestibular Ocular; Postural Balance
MeSH Terms: conditions — Vestibular Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- control (No Intervention): Control without vestibular stimulation
- Bilateral areflexia (No Intervention): Patient with vestibular bilateral areflexia
- Areflexia controls (No Intervention): Controls for patients with vestibular bilateral areflexia, matched in sex and age
- vestibular stimulation (Experimental): Subjects submitted to vestibular stimulation in order to improve circadian rhythms
  Interventions: Behavioral: vestibular stimulation

INTERVENTIONS:
Behavioral: vestibular stimulation — Physical activity and vestibular stimulation will be used in order to improve circadian rhythms
  Arms: vestibular stimulation

SUMMARY:
The purpose of this study is to study the relationship between the vestibular system and chronobiology

DETAILED DESCRIPTION:
The purpose of this study is to study the relationship between the vestibular system and chronobiology.

Two parts will be performed. In the first one patients with bilateral vestibular areflexia will be compared to control subjects.

In the second the effect of vestibular stimulation on circadian rhythms will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* No treatment changing vigilance/wakefulness
* Moderate caffein uptake (2 to 3 cups a day)
* Moderate smoker (5 cigarettes a day)
* Regular sleeping habits

Exclusion Criteria:

* Sleeping duration <6 hours or >9 hours
* Night workers
* Pregnancy
* Sleep or wakefulness disorders
* Progressive neurodegenerative disorders
* Progressive psychiatric disorders
* Thyroid disease
* Type 1 diabetes
* Not able to practice physical activity
* Drug or alcohol addiction during the last 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Measurements of vestibular reflexes (ocular and spinal) and circadian rhythms of biological functions. | 3 years
  Gain of vestibular ocular reflex Amplitude of vestibular spinal reflex Amplitude and phase of temperature circardian rhythms

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Denise, MD, PhD, Principal Investigator — University Hospital of Caen
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France